CLINICAL TRIAL: NCT00210782
Title: A Double-blind Trial Comparing the Efficacy, Tolerability and Safety of Monotherapy Topiramate Versus Phenytoin in Subjects With Seizures Indicative of New Onset Epilepsy
Brief Title: A Comparison of the Effectiveness and Safety of Topiramate and Phenytoin in Patients With New Onset Epilepsy Requiring Rapid Initiation of Antiepileptic Drug Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004663
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Epilepsy
Keywords: epilepsy; seizures; epileptic seizures; complex partial seizures; generalized tonic-clonic seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Topiramate; Phenytoin

INTERVENTIONS:
Drug: topiramate, phenytoin

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of two treatment regimens, topiramate as compared to phenytoin, in preventing seizures in patients with new-onset epilepsy who require rapid initiation of antiepileptic drug therapy. Reasons for requiring rapid initiation of treatment, rather than slowly increasing an antiepileptic drug to an effective dose, may include severe or frequent seizures, or high risk to the patient of recurrent seizures.

DETAILED DESCRIPTION:
In this study, patients who have recently been diagnosed with epilepsy and who require rapid initiation of treatment will be randomized to receive either phenytoin or topiramate. Patients have an equal chance of receiving either medication. Phenytoin and topiramate have been approved by the FDA for treatment of epilepsy. The first phase of this study (lasting 28 days) is double-blind, meaning that neither the patient or the physician know which medication the patient is receiving. Phenytoin will be used according to the dosing recommendation in the package insert. Patients randomized into the phenytoin arm of this study, will receive a dose on day 1 of 1000mg phenytoin (given in 3 divided doses), an initiation dose recommended in the product labeling. This will be followed by 300mg of phenytoin on each subsequent day. Patients randomized into the topiramate arm of this study will receive 100mg of topiramate on day 1 and then continue to receive 100mg on each subsequent day. This is a relatively rapid initiation schedule of topiramate, but it is anticipated that it will be well tolerated and represents an appropriate regimen for comparison to patients in the phenytoin arm of the study. Patients will be carefully monitored for primary generalized tonic clonic seizures or complex partial onset seizures (two distinct epileptic seizure types) during the 28-day double-blind evaluation period of the trial. If a patient experiences a seizure during this 28 day period, they will either be taken out of the study, or be offered the option to receive a higher dose of topiramate in an open-label fashion. Open-label means that the patient and the physician will know what medication and what dose of the medication the patient is taking. All patients who do not experience a seizure during the 28 day period will be offered to receive open-label topiramate for an additional 12 weeks. The study hypothesis is that the proportion of patients who do not have a seizure within the 28 day double blind phase of the study will not differ between the 2 treatment groups. Topiramate 100 milligrams a day by mouth for 4 weeks; phenytoin 1000 milligrams to start, decreased to 300 milligrams a day by mouth for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Seizures indicative of new-onset epilepsy (or epilepsy relapse) of untreated epilepsy
* at least one but not more than 20 unprovoked seizures within past 3 months
* weighing more than 110 pounds
* considered to be a good candidate for rapid initiation of anti-seizure medication
* able to swallow a tablet whole (without crushing it).

Exclusion Criteria:

* Not having taken anti-seizure medications within the past 30 days
* no provoking factors for seizures (presence of alcohol withdrawal, drug intoxication, acute meningitis or encephalitis, acute head injury or stroke, acute hypoxic/ischemic encephalopathy, or brain tumor)
* no presence of active liver disease or serious kidney disease
* not pregnant or breast-feeding
* not using birth control.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2004-06; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome parameter is the time to first seizure during the double blind phase of the study. The statistical evaluation will analyze if there is a significant difference in the proportion of patients being seizure free between both medications.

SECONDARY OUTCOMES:
Effect of sex, age, baseline weight, baseline seizure type, and duration since first diagnosis of epilepsy on the time to seizure.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Ramsay E, Faught E, Krumholz A, Naritoku D, Privitera M, Schwarzman L, Mao L, Wiegand F, Hulihan J; CAPSS-272 Study Group. Efficacy, tolerability, and safety of rapid initiation of topiramate versus phenytoin in patients with new-onset epilepsy: a randomized double-blind clinical trial. Epilepsia. 2010 Oct;51(10):1970-7. doi: 10.1111/j.1528-1167.2010.02670.x. PMID 20633037
- See also: Topiramate vs. Phenytoin in New Onset Epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=616&filename=CR004663_CSR.pdf